CLINICAL TRIAL: NCT05377515
Title: Evaluation of Visual Outcomes in Patients With Complex Corneas Implanted With the IC-8 IOL
Status: Completed | Type: Observational
Sponsor: AcuFocus, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IC8-303-EXPA
Record Dates: First submitted 2022-05-12; First posted 2022-05-17 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Cataract; Presbyopia; Irregular; Contour of Cornea
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IC-8 IOL Group: Visual outcomes in patients previously contralaterally implanted with the IC-8 IOL will be evaluated.

SUMMARY:
The purpose of this study is to evaluate visual outcomes in patients with complex corneas who have been previously implanted with the IC-8 IOL after cataract removal.

DETAILED DESCRIPTION:
This will be a prospective, non-randomized, single-arm, single-visit, single-center, clinical study in up to 40 patients previously contralaterally implanted with the IC-8 IOL at one clinical site in Singapore.

The purpose of this study is to to evaluate visual outcomes in patients with complex corneas who have been previously implanted with the IC-8 IOL after cataract removal. The co-primary study endpoints are monocular uncorrected distance, intermediate, near visual acuities.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum 22 years of age;
2. Able to comprehend and have signed a statement of informed consent;
3. Availability, willingness, ability and sufficient cognitive awareness to comply with examination procedures and study visit(s);
4. Having complex corneas prior to cataract surgery;
5. Previous cataract surgery and IC-8 IOL implantation in the eye (implanted for 3 months or longer prior to study participation).

Exclusion Criteria:

1. Baseline visual acuity worse than 20/25 BCDVA in either eye;
2. Presence of ocular abnormalities or conditions other than corneal irregularities that could confound the study outcome(s), such as:

   1. Strabismus or amblyopia
   2. Retinal or macular abnormalities
   3. Recurrent and/or persistent ocular inflammation
   4. Known pathology that may affect visual acuity to a level worse than 20/25 BCDVA
3. Previous intraocular surgery, except cataract surgery, pterygium surgery, or corneal procedures (other than corneal-cross linking);
4. Previous corneal cross-linking procedure with any corneal haze;
5. Conditions requiring planned ocular surgical intervention, except Nd:YAG capsulotomy;
6. Severe dry eye or other conditions (such as hormonal fluctuations) that could lead to unstable refraction and/or visual acuity measurements or eye discomfort even with ocular lubricants or dry eye medication;
7. Patient is pregnant or nursing.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients for this study will be recruited from patients with complex corneas who have been previously implanted with the IC-8 IOL after cataract removal. Anticipated study sample size of up to 40 patients will be evaluated.
  Patients will be screened for eligibility, and an informed consent will be obtained from those who meet the screening criteria and are interested in participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Monocular UCDVA | 3 Months
  0.3 logMAR or better
Monocular UCIVA | 3 Months
  0.3 logMAR or better
Monocular UCNVA | 3 Months
  not worse than 0.3 logMAR

CONTACTS AND LOCATIONS:
Overall Officials: Magda Michna, Ph.D., Study Director — AcuFocus, Inc.
Locations (1):
- Singapore Eye Research Institute / Singapore National Eye Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No